CLINICAL TRIAL: NCT05391906
Title: Intravoxel Incoherent Motion (IVIM) Magnetic Resonance Imaging in Multiple Sclerosis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Tiffany So, Clinical Assistant Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TiffanySo
Record Dates: First submitted 2022-05-03; First posted 2022-05-26 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intravoxel Incoherent Motion(IVIM) MRI (Experimental): Intravoxel incoherent motion (IVIM) is based on diffusion-weighted imaging (DWI)
  Interventions: Other: Diffusion-weighted magnetic resonance imaging

INTERVENTIONS:
Other: Diffusion-weighted magnetic resonance imaging — Diffusion-weighted magnetic resonance imaging
  Other Names: Diffusion-weighted magnetic resonance imaging uses the diffusion of water molecules to generate contrast in MR images.

SUMMARY:
Intravoxel incoherent motion (IVIM) is technique based on diffusion-weighted imaging (DWI). In this study, the investigators evaluate the use of IVIM in patients with Multiple Sclerosis.

DETAILED DESCRIPTION:
Intravoxel incoherent motion (IVIM) is technique based on diffusion-weighted imaging (DWI), it is achieved through an MRI acquisition with multiple small b value to extract perfusion data. It has been shown to be a promising technique in evaluation of many brain conditions. This study seeks to assess intravoxel incoherent motion (IVIM) parameters in characterizing plaques and specific tissues in multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are 18 years or older.
2. Relapsing-remitting MS diagnosed as per Macdonald criteria

Exclusion Criteria:

1. Contraindication to MRI. For example, metal implantation in the body, claustrophobia and pregnancy.
2. Patients who are unable to tolerate the scans without moving the head as a result of symptoms such as tremor, spasticity, involuntary movements and spasms, cognitive impairment, coughing, and shortness of breath.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2026-12-20 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
IVIM parameters (including ADC,D,D*,f) in Multiple Sclerosis brain regions. | Up to 2 months
  Primary Outcome Measure:
  1. IVIM parameters (including ADC,D,D*,f) in Multiple Sclerosis brain regions. The parameters are calculated based on a IVIM model bi-exponential model represented by: S(b)/S(0)=f ×exp(-bD*)+ (1-f)×exp(-bD), and the mono-exponential model for ADC calculation as represented by: S(b)/S(0)=exp(-bADC), where S(b) and S (0) are the MRI signal intensities at a given b value and b = 0, respectively.
  ADC: apparent diffusion coefficient. ADC is expressed in units of mm2/s.
  f: the perfusion or (micro) vascular volume fraction which depends on capillary geometry and blood velocity. f is expressed in units of mm2/s.
  D*: pseudo diffusion coefficient that resembles the perfusion related incoherent microcirculation. D* is expressed in units of mm2/s.
  D: pure diffusion coefficient which is related to pure molecular diffusion. D is expressed in units of mm2/s.

CONTACTS AND LOCATIONS:
Locations (1):
- CUHK, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No